CLINICAL TRIAL: NCT04760470
Title: Technology-assisted Upper Extremity Rehabilitation in Subjects with Incomplete Cervical Spinal Cord Injury - Randomized Controlled Crossover Trial
Brief Title: Technology-assisted Upper Extremity Rehabilitation in Subjects with Incomplete Cervical Spinal Cord Injury
Acronym: T-ARSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: The Finnish Association of People with Physical Disabilities (Other); Helsinki University Central Hospital (Other); Validia Rehabilitation (Unknown)
Responsible Party: Principal Investigator, Joonas Poutanen, Principal investigator, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01012021
Record Dates: First submitted 2021-02-06; First posted 2021-02-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Technology-assisted upper extremity rehabilitation (Experimental): Technology-assisted upper extremity rehabilitation.
  Interventions: Other: Technology-assisted upper extremity rehabilitation
- Wait list control (No Intervention): Continue their normal lives.

INTERVENTIONS:
Other: Technology-assisted upper extremity rehabilitation — Subjects get 6 weeks of technology-assisted upper extremity rehabilitation
  Arms: Technology-assisted upper extremity rehabilitation

SUMMARY:
The aim of the study is to investigate the effects of 6 weeks of technological-assisted rehabilitation on function of upper extremity and hand in subjects with incomplete cervical spinal cord injury.

DETAILED DESCRIPTION:
In this crossover study, persons with motor incomplete cervical (C2-C8) spinal cord injury (AIS C-D) will be recruited from the Hospital District of Helsinki and Uusimaa. In the first period of the crossover study, other part of the participants will get technological-assisted upper extremity rehabilitation, while the other part of the participants continue their normal lives. The first period is followed by 4-week wash-out period. In the second period, roles of the participants will be switched. The rehabilitation phase lasts for 6 weeks with 3 weekly sessions, each therapy session including at least 30 minutes of technological-assisted upper extremity rehabilitation. Rehabilitation includes passive, active and resistance exercises, and will be carried out by using AMADEO, PABLO and/or DIEGO devices made by Tyromotion.

ELIGIBILITY:
Inclusion Criteria:

* incomplete motor spinal cord injury (AIS C-D)
* injury level C2-C8
* time since injury from 1 to 5 years
* to be able to sit
* motivation and ability to participate in intensive rehabilitation 3 times per week for 6 week period.

Exclusion Criteria:

* participation in other exercise study or technological-assisted upper extremity study
* unlikely completion of intervention and participation in follow up
* injuries that prevent training
* weak tolerance of intense training
* severe joint movement restriction or instability
* irreversible muscle contractures
* grade 4 on Modified Ashworth Scale in glenohumeral, elbow, wrist and finger joints
* recent significant forearm or hand injuries
* memory disorder
* orthopedic, rheumatic or neurological diseases (other than spinal cord injury) that prevent training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | 6 weeks,16 weeks, and 6 months
  Maximum score is 114 (on a scale from 0 to 114) as the higher score indicate better upper extremity functioning.
Goal Attainment Scaling (GAS) | 6 weeks or 16 weeks
  A method to evaluate rehabilitation effects. A 5-point scale ranging from -2 to 2. Zero represents expected level of performance after rehabilitation, +1 more than expected, and +2 much more than expected. Respectively, -1 means less than expected and -2 much less than expected.

SECONDARY OUTCOMES:
American Spinal Injury Association - Upper Extremity Motor Scores (ASIA-UEMS) | 6 weeks,16 weeks, and 6 months
  Maximum score is 50 (on a scale from 0 to 50) as the higher score indicate better motor functioning in upper extremities.
Grip strength | 6 weeks,16 weeks, and 6 months
  Measured with Jamar-dynamometer
Pinch strength | 6 weeks,16 weeks, and 6 months
  Measured with
Upper extremity active range of motion | 6 weeks,16 weeks, and 6 months
  Measured with goniometer
Spinal Cord Independence Measure - Self Report (SCIM-SR) | 6 weeks,16 weeks, and 6 months
  Maximum score is 100 (on a scale from 0 to 100) as the higher score indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sinikka Hiekkala, PhD, Study Director — The Finnish Association of People with Physical Disabilities
Locations (1):
- Validia Rehabilitation, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No